CLINICAL TRIAL: NCT02813226
Title: Assessment of New Molecular Imaging Strategies for Prostate Cancer: Predictive Value of Established and Novel Positron Emission Tomography (PET) Radiotracers in Castration-Resistant Prostate Cancer
Brief Title: Assessment of New Molecular Imaging Strategies for Prostate Cancer
Acronym: MISTER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OCOG-2016-MISTER
Record Dates: First submitted 2016-06-22; First posted 2016-06-24 (Estimated); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Prostate Cancer
Keywords: castration-resistant; molecular imaging; abiraterone acetate; enzalutamide; metabolic response
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Molecular Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Imaging (Other): Molecular Imaging
  Interventions: Other: Molecular Imaging

INTERVENTIONS:
Other: Molecular Imaging — Baseline and follow-up FDG PET-CT and DCFPyL PET-CT

SUMMARY:
In this study 30 men, with advanced metastatic Castration-Resistant Prostate Cancer (CRPC) planned to have hormonal treatment, will undergo conventional imaging and functional imaging prior to treatment and post treatment to determine if changes in imaging results will be prognostic of outcome. Patients will have a clinical follow-up every 3 months post randomization for one year and followed for survival at Years 2 and 3.

DETAILED DESCRIPTION:
In this study 30 men, with advanced metastatic CRPC intended to have abiraterone acetate or enzalutamide hormonal treatment will undergo conventional imaging including a 99mTc-Methyl diphosphonate (MDP) bone scan and Computed Tomography (CT) of the abdomen and pelvis, and functional imaging with 18F-fluorodeoxyglucose (FDG) PET-CT and 2-(3-(1-carboxy-5-[(6-[18F]fluoro-pyridine-3-carbonyl)-amino]-pentyl)-ureido)-pentanedioic acid (18F-DCFPyL) PET-CT one to four weeks prior to hormonal treatment and approximately 10 weeks post hormonal treatment.

Prostate Specific Antigen (PSA) will also be obtained at baseline and every three months in the first year. Baseline imaging of disease and changes between baseline and follow-up imaging on 18F-FDG PET-CT and 18F-DCFPyL PET-CT will be compared with standard of care imaging (99mTc-MDP bone scan and CT of the abdomen/pelvis) as well as with clinical evaluation including response to therapy and progression of disease.

This information could be used by clinicians to guide androgen receptor (AR) - targeted therapy. Patients will have a clinical follow-up every 3 months post randomization for one year and will be followed for survival at Years 2 and 3.

ELIGIBILITY:
Inclusion Criteria:

1. Objectively documented metastatic prostate cancer progression with either of the following:

   * At least one rising PSA over a minimum of one week interval within six weeks of study registration, or
   * Radiographic progression in soft tissue and/or bone within six weeks of study registration
2. Ongoing androgen deprivation therapy with serum testosterone <50 ng/dL (<1.7 nmol/L).
3. Planned to start abiraterone acetate or enzalutamide.

Exclusion Criteria:

1. Age < 18 years.
2. Eastern Cooperative Oncology Group (ECOG) performance status >2.
3. Planned to receive palliative radiotherapy within the next 12 weeks.
4. Hemoglobin < 90 g/L independent of transfusion.
5. Platelet count < 50 x 10^9 / L.
6. Serum albumin < 30 g/L.
7. Serum creatinine > 1.5 x Upper Limit of Normal (ULN) or a calculated creatinine clearance <30 L/min.
8. Contraindications to FDG.
9. Inability to lie supine for imaging with PET-CT.
10. Inability to undergo CT due to known allergy to contrast.
11. Inadequate hepatic function: (i) Bilirubin >1.5 x ULN, and (ii) Serum glutamic oxaloacetic transaminase (SGOT) >3 x ULN
12. Inability to complete the study or required follow-up

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2021-12-17 (Actual)

PRIMARY OUTCOMES:
Functional imaging metabolic response contrasted with conventional imaging response | 10 weeks
  Percent change of the average maximum standardized uptake value (SUVmax) of target lesions in contrast with conventional imaging soft tissue and bone response between the baseline scans and the Week 10 scans.

SECONDARY OUTCOMES:
Functional imaging response | 10 weeks
  The percent change in the SUVmax of the most intensely FDG/DCFPyL avid lesion relative to Baseline.
Radiological progression free survival. | 3 years
  The time from registration to the first date of radiographic disease progression in bone or soft tissue or to the date of death
Prostate specific antigen (PSA) response | 3 years
  The time from registration to the date of PSA progression
Progressive Disease (example change in treatment, skeletal related event) | 3 years
  The time from registration to initiation of anti-cancer intervention or death from any cause.
Overall Survival | 3 years
  The time from registration to the date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Zukotynski, Principal Investigator — Hamilton Health Sciences Corporation; Eric Winquist, Principal Investigator — London Health Sciences Centre
Locations (3):
- Canada (3):
  - Juravinski Hospital and Cancer Centre, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Sunnybrook-Odette Cancer Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No